CLINICAL TRIAL: NCT05276362
Title: Study Watch Sleep Metric Performance Characterization Study
Status: Completed | Type: Observational
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 103845
Record Dates: First submitted 2022-02-25; First posted 2022-03-11 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Sleep; Obstructive Sleep Apnea; Insomnia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- Typical Sleepers: This will be a single arm study of approximately 70 typical sleepers that will wear the Study Watch(es) and Actiwatch for one night in a sleep laboratory.
  Interventions: Device: Study Watch; Device: Actiwatch
- Sleepers with Elevated Insomnia Symptoms: This will be a single arm study of at least 15 participants with elevated insomnia symptoms that will wear the Study Watch(es) and Actiwatch for one night in a sleep laboratory.
  Interventions: Device: Study Watch; Device: Actiwatch
- Sleepers withObstructive Sleep Apnea Sleepers: This will be a single arm study of at least 15 participants with obstructive sleep apnea that will wear the Study Watch(es) and Actiwatch for one night in a sleep laboratory.
  Interventions: Device: Study Watch; Device: Actiwatch

INTERVENTIONS:
Device: Study Watch — The Study Watch is an investigational wrist worn wearable device made with biocompatible contact materials containing various sensors capable of continuous recording of physiological, activity, and environmental data.
Device: Actiwatch — The Actiwatch is a wrist worn activity device designed to collect general activity and sleep information. This device received 510(k) clearance from the FDA as a wearable medical data collection device for research and clinical use.

SUMMARY:
This is a multi-center, single-arm, prospective performance evaluation study designed to assess performance of sleep metrics calculated from sensor data that is collected from two versions of the Verily Study Watch as compared to polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 18 and ≤ 80 years old
* Participant understands the study requirements and is able and willing to provide written informed consent
* Participant is without significant limitation in ability to participate in the study, in the opinion of the investigator
* Participant belongs to one of the following participant groups as determined by screening questionnaires:

  * Typical sleepers (i.e., STOP-Bang score of 0-2 or OSA50 < 5, Insomnia Severity Index (ISI) < 8, and Epworth Sleepiness Scale (ESS) < 10), and no evidences of sleep-disordered breathing at the PSG evaluation
  * Insomnia sleepers (i.e., ISI > 10 and PSG AHI < 5)
  * Sleep apnea sleepers (i.e., STOP-Bang score of 3-8 or OSA50 ≥ 5) or moderate to severe obstructive sleep apnea (PSG AHI ≥5))
* Participant has agreed to abstain from caffeine, nicotine, alcohol, and cannabis products for 8 hours prior to the In-Lab Screening Visit and until the visit is completed

  * Exception - unless the participant use of product has approval from the Principal Investigator
* Participant has agreed to abstain from OTC or PRN medications that are not regularly used on a daily basis and may affect sleep/wakefulness for 24 hours prior to the In-Lab Overnight Visit and during the study visit

  * Exception - unless the participant uses OTC or PRN medication on a routine basis and has approval from the Principal Investigator

Exclusion Criteria: Conditions based on self-report of having been told by a doctor of a formal diagnosis

* Presence of any of the following diagnosed sleep, medical, or psychiatric disorders:

  * Sleep

    * Narcolepsy
    * Restless leg syndrome
    * Circadian rhythm sleep disorder
    * Periodic Limb Movement Disorder
    * REM Sleep behavior disorder
  * Medical

    * Epilepsy or other seizure disorder
    * Renal failure or chronic kidney disease
    * Acute or chronic infection that may interfere with the study
    * Movement neurological disorder that impairs movement or autonomic stability (e.g. Parkinson's disease, Huntington's disease)
    * Cardiopulmonary diseases (e.g. heart failure, chronic obstructive pulmonary disease, ventilatory disorders)
    * Persistent arrhythmias and dysrhythmias
    * Severe neuromuscular disease (e.g. Amyotrophic lateral sclerosis [ALS])
  * Psychiatric

    * Severe significant mood disorder (e.g. depression, bipolar disorder)
    * Substance use disorder
* Participant uses supplemental oxygen during the day or night
* Participant is unwilling to cease use of CPAP or oral appliance for sleep-disordered breathing during the In-Lab Overnight Visit; or cessation is deemed to be of substantial risk in the opinion of the Principal Investigator
* Women who are pregnant, lactating, or breastfeeding
* Participant takes prescription stimulants, sedatives, opioids, alpha blockers, short acting nitrates, or any other medication that, in the opinion of the Principal Investigator and study team, impacts their sleep behavior
* Use of any sleep medications (over-the-counter or prescription) in the previous 24 hours for Typical Sleepers
* Participant has a cardiac pacemaker, implantable defibrillator, medical pump, or other implantable medical electronic device
* Participant has Shift Work Sleep Disorder (SWSD) or is a night-shift worker
* Participant has traveled >3 time zone within two weeks prior to study
* Participant is not fluent at reading and speaking English
* Participant is deemed not to be a candidate for the study, in the opinion of the Principal Investigator
* Known severe allergy to nickel or metal jewelry
* Open injury or rash where the study device or comparator will be worn
* Known severe allergy to polyester, nylon, or spandex material
* Enrolled participants who meet exclusion criteria after PSG, upon confirmation with the principal investigator and study team, will be discontinued and excluded from primary analyses.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Complete datasets will be collected on approximately 70 typical sleepers, at least 15 participants with Obstructive Sleep Apnea (OSA), and at least 15 participants with elevated insomnia symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of sleep/wake detection - Sensitivity and Specificity | 1 night
  Accuracy of sleep/wake detection will be reported on 30 second epochs from lights off to lights on in typical sleepers.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Nelson, PhD, Study Director — Verily Life Sciences
Locations (1):
- SRI International, Menlo Park, California, United States

REFERENCES:
- [Derived] Saeb S, Nelson BW, Barman P, Verma N, Allen H, de Zambotti M, Baker FC, Arra N, Sridhar N, Sullivan SS, Plowman S, Rainaldi E, Kapur R, Shin S. Performance of the Verily Study Watch for measuring sleep compared to polysomnography. Front Sleep. 2024 Dec 13;3:1481878. doi: 10.3389/frsle.2024.1481878. eCollection 2024. PMID 41424491